CLINICAL TRIAL: NCT05626816
Title: Short-term Genital Nerve Stimulation to Modulate Anorectal Reflex Activity in Neurogenic Bowel Dysfunction in Individuals Living With Spinal Cord Injury
Brief Title: Acute Genital Nerve Stimulation for Neurogenic Bowel Dysfunction in Individuals Living With Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: VA of Northeast Ohio Health System (Unknown); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Hoey, Associate Professor, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000105; CDMRP-SC210121P1 (Other Grant/Funding Number: Department of Defense CDMRP SCIRP); CDMRP-SC210121 (Other Grant/Funding Number: Department of Defense CDMRP SCIRP)
Record Dates: First submitted 2022-10-19; First posted 2022-11-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Fecal Incontinence
Keywords: bowel; spinal cord injury; electrical stimulation; anorectal manometry; incontinence; tetraplegia; paraplegia; paralysis
MeSH Terms: conditions — Fecal Incontinence; Spinal Cord Injuries; Quadriplegia; Paraplegia; Paralysis

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention, but randomization will determine the order of presentation of sham and effective stimulation to ensure blinding of the participant.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- All interventions, Sham applied first (Experimental): These participants will have all interventions applied, but will be randomly designated to have sham stimulation applied before effective stimulation. This will balance any issue with order of presentation of multiple stimulation sessions.
  Interventions: Device: Genital Nerve Stimulation; Diagnostic Test: Clinical exam; Diagnostic Test: Collection of SCI common data elements; Diagnostic Test: Bowel function survey completion; Diagnostic Test: International Standard for Neurological Classification of SCI (ISNCSCI); Diagnostic Test: Response to genital nerve stimulation (GNS); Diagnostic Test: Anorectal Manometry testing (ARM)
- All interventions, effective stim applied first (Experimental): These participants will have all interventions applied, but will be randomly designated to have effective stimulation applied before sham stimulation. This will balance any issue with order of presentation of multiple stimulation sessions.
  Interventions: Device: Genital Nerve Stimulation; Diagnostic Test: Clinical exam; Diagnostic Test: Collection of SCI common data elements; Diagnostic Test: Bowel function survey completion; Diagnostic Test: International Standard for Neurological Classification of SCI (ISNCSCI); Diagnostic Test: Response to genital nerve stimulation (GNS); Diagnostic Test: Anorectal Manometry testing (ARM)

INTERVENTIONS:
Device: Genital Nerve Stimulation — Electrical stimulation applied to the genital nerve with surface electrodes using an off the shelf TENS unit (Ultima Plus). First, an amplitude threshold for the pudendo-anal reflex responses will be determined. Then, sham (1-2 Hz) and effective stimulation (20 Hz) will be briefly applied to record responses. Then, stimulation will be applied in random presentation order to record any changes in anorectal manometry outcomes due to both sham and effective stimulation.
Diagnostic Test: Clinical exam — Examination by physician determines the presence of pelvic reflexes (pudendo-anal and bulbocavernosus) which are essential for GNS to have an effect.
Diagnostic Test: Collection of SCI common data elements — Data regarding participant demographics, history of injury, and medical history will be collected.
Diagnostic Test: Bowel function survey completion — Two surveys will be conducted to assess the bowel function of the participant. The International SCI Bowel Function Basic Data Set (ISCI BF BDS v2.1) and the SCI Qulaity of Life Bowel Management Difficulties (SCI-QoL BMD) survey scales collect data on overall bowel function and how any difficulties impact the participants quality of life.
Diagnostic Test: International Standard for Neurological Classification of SCI (ISNCSCI) — The physician will conduct the ISNCSCI to determine the level and severity of injury to the spinal cord. This is done by determining the ability to detect light touch and pinprick stimulation. Outcomes will be a Spinal Injury Association Impairment Scale (AIS) grade of A-D.
Diagnostic Test: Response to genital nerve stimulation (GNS) — GNS will be applied to determine if there is a response in the participant. If the participant has no response to the stimulation they will be excluded from the second visit as it is dependent on the ability to respond to GNS.
Diagnostic Test: Anorectal Manometry testing (ARM) — The participant will be instrumented for ARM testing. This requires a special balloon catheter to be inserted into the anus and secured, surface electrode pads being applied to the anal sphincter, and electrode pads being applied to the genital nerve stimulation sites.
  Once instrumented, the participant will be tested with the London Classification procedure. This procedure asks the participant to perform several actions (squeeze to withhold a bowel movement, push to have a bowel movement, and cough) as well as inflating the balloon on the catheter to determine reflex thresholds (RAIR, retroanal inhibitory reflex which relaxes the anal sphincter in response to rectal distension) and sensory thresholds (first senstation,

SUMMARY:
Bowel issues occur in nearly all people after spinal cord injury (SCI) and one major complication is fecal incontinence (accidents). This complication has been repeatedly highlighted by people living with SCI as particularly life-limiting and in need of more options for interventions. This study will test the effect of genital nerve stimulation (GNS), with non-invasive electrodes, on the activity of the anus and rectum of persons after SCI. Recording anorectal manometry (ARM) endpoints tells us the function of those tissues and our study design (ARM without stim, ARM with stim, ARM without stim) will allow us to conclude the GNS effect and whether it is likely to reduce fecal incontinence. The study will also collect medical, demographic, and bowel related functional information. The combination of all of these data should help predict who will respond to stimulation, what will happen when stimulation is applied, and if that stimulation is likely to provide an improvement in fecal continence for people living with SCI.

DETAILED DESCRIPTION:
Time commitment: A person who participates in this study will have the option of coming in for one or two visits (for a total of about 7.5 hours). Descriptions below will separate the research activities into two visits for clarity.

Minimizing barriers to participation:

1. - If you live in the region (Cuyahoga, Lorain, Medina, Lake, or Geauga counties of Ohio) and need assistance with transportation to get to and from the research site for a visit, the study team will make these arrangements at no cost to you. If you live outside of the region, the study team will reimburse your transportation expenses up to a maximum of $556 per visit.
2. - If you live a distance away from the research site for which it would be easier for you to spend the night closer for a research visit, accessible lodging is available at the Zubizarreta House. This house is right next door to the MetroHealth Rehabilitation Institute and is designed for people with spinal cord injuries. The overnight stay will be provided at no cost to you, but if you need a caregiver to stay with you that is your responsibility.

Visit 1 (screening): When a person decides to participate in the study they will be scheduled to come in for a screening visit. During this visit they will: provide informed consent to participate, participate in the initial screening exams, and have genital nerve stimulation (GNS) applied briefly to determine if the nerve responds to electrical stimulation.

If a person completes the screening procedures and qualifies for the study they will be invited back to complete the manometry visit.

Visit 2 (manometry):

1. - Preparation: the participant will be asked to complete their typical bowel program the night before their manometry visit is scheduled. There are no restrictions on medications, eating, or drinking prior to the visit.
2. - Instrumentation: the participant will have the study instrumentation applied.
3. - Testing procedures with ARM and GNS: The London classification protocol will be used to assess ano-rectal function. This procedure uses a short (~12 minutes) procedure of actions to determine how the anus and rectum are functioning.

Overall design: GNS and the London classification system will be used to assess bowel function in two different states, with stimulation and without stimulation. This will be applied in the order of no stimulation (condition A), stimulation (condition B), no stimulation (condition A repeated).

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI
* Minimum 6 months post-injury
* Aged 18 years or older
* Neurological level of injury T12 or higher AIS grade A-D defined by ISNCSCI
* Response to genital nerve stimulation upon screening
* Able to understand and provide informed consent

Exclusion Criteria:

* Currently enrolled in another functional electrical stimulation (FES) research trial
* Females who are pregnant or planning to become pregnant during the trial
* Presence of cardiac pacemaker, implanted defibrillator or other implanted FES device if, upon clinical exam, it may have an interaction with GNS.
* In the judgement of the PI or Co-Investigators, presence of medical complications that may interfere with the execution of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ARM outcome - Rectal wall tension | Up to three weeks after enrollment
  When an organ relaxes during filling it is called compliance and is characteristic of the rectum and bladder. This allows the organ to hold more material and therefore have a larger void when emptying. After SCI, organs that have had their control systems damaged become spastic and hyperreflexive which leads to smaller volumes and incontinence issues in both bladder and bowel function.
  By inflating the ARM balloon with air we can slightly distend the rectum and measure the pressure (cmH20) to determine compliance. If the pressure stays the same after inflating the balloon then the rectum has relaxed and it is a measure of compliance. Rectal wall tension will be inferred from this response and abnormal tension will be apparent by reduced compliance (pressure increases when balloon volume increases).
  This measure will be recorded with and without stimulation.
ARM outcome - Anal sphincter function | Up to three weeks after enrollment
  Circumferential sensors on the ARM balloon catheter will detect pressure changes (cmH20) in the anal sphincter during cough, push, squeeze, and rest. Anal sphincter function will be assessed with and without stimulation.
ARM outcome - Rectoanal reflex activity (RAIR) | Up to three weeks after enrollment
  Air will be infused into the ARM balloon to distend the rectum. When the rectum is distended the anal sphincter relaxes (rectoanal inhibitory reflex) and the amount of air required to elicit the reflex (cc) will be assessed with and without stimulation.
ARM outcome - Rectal sensation | Up to three weeks after enrollment
  Air is infused (50 ml steps) into the ARM balloon until the participant reports: first sensation, urge to defecate, maximum tolerable sensation. The volume of air (cc) is recorded for each sensory event with and without stimulation.
ARM outcome - Presence of hyper reflexive rectal contractions | Up to three weeks after enrollment
  After SCI the rectum become hyperreflexive and spastic. A major cause of fecal incontinence after injury is the result of these reflexive contractions and the inability to contract the external sphincter to maintain continence. This combination causes the rectum to expel small amounts of stool rather than storing the material for a larger bowel movement.
  We will quantify the rectal pressure traces for reflexive contractions and measure their frequency (Hz or count/minute, whichever is most appropriate). Reflexive contractions will be steep increases in rectal pressure while at rest or during distension (sensation and RAIR testing). Measurements will be collected with and without stimulation and compared.

SECONDARY OUTCOMES:
SCI-QOL Bowel Management Difficulties (SCI-QOL BMD) | During enrollment, up to one week
  A survey on bowel management difficulties and the effect of those complications on the participants quality of life will be conducted and data collected by study staff. Answers are chosen from a 5-point Likert scale from 1 (never/not at all) to 5 (always/very much) and higher scores represent greater difficulty managing bowel complications.
International SCI Bowel Function Basic Dataset Version 2.1 (ISCI BF BDS) | During enrollment, up to one week
  A survey on bowel function after SCI will be conducted and data collected by study staff. The instrument is on a scale from 0-45 with higher scores indicating greater dysfunction.
International Standards of Neurological Classification of SCI (ISNCSCI) | During enrollment, up to one week
  This is a standard assessment tool to determine level and severity of injury by the American Spinal Injury Association. The test uses pin prick and light touch to determine motor and sensory capability along the body. At the end of the test the participant will have information on their level (i.e. T8) and severity (grade A-D, with A being motor and sensory complete injury). These endpoints overlap with the clinical exam outcomes and will only be conducted once. Therefore, the ISNCSCI is being conducted in the context of the clinical exam endpoints below.
SCI Common Data Elements - Medical history | During enrollment, up to one week
  Data will be collected regarding body system categories (constitutional symptoms, eyes, ears/nose/mouth/throat, cardiovascular, respiratory, gastrointestinal, genitourinary, musculoskeletal, integumentary, neurological, psychiatric, endocrine, hematologic/lymphatic, and allergic/immunologic) including start date, end date, and ongoing status.
SCI Common Data Elements - History of injury | During enrollment, up to one week
  Data regarding the injury etiology and time frame will be collected from the participant.
SCI Common Data Elements - Demographics | During enrollment, up to one week
  Data regarding the participants' gender, birth date, race, ethnicity, marital status, number of members in household, area of residence, number of years of education, and primary occupation.
Clinical exam - abdominal exam | During enrollment, up to one week
  An SCI-specialized clinician will assess the participant in regard to abdominal health. This data will be incorporated into a clinical characterization of bowel dysfunction.
Clinical exam - Evaluation of sacral reflexes | During enrollment, up to one week
  An SCI-specialized clinician will assess the participant in regard to the integrity of the sacral reflexes. These include the pudendo-anal reflex (PA) and bulbocavernosus (BC) reflexes that are critical for responding to the genital nerve stimulation.
Clinical exam - Anal sphincter tone | During enrollment, up to one week
  An SCI-specialized clinician will assess the participant in regard to anal sphincter tone. After injury the external anal sphincter is either spastic (tightly closed and difficult to relax) or flaccid (completely lax and does not contract) based on the level of injury. If the damage to the spinal cord is at the level of the sacrum (just above the tailbone area) it will cause a flaccid phenotype and indicates damage to the reflex pathways necessary for the experiment.
Clinical exam - Sensation | During enrollment, up to one week
  An SCI-specialized clinician will assess the participant in regard to areas of the body that have sensation. This data is incorporated in the ISNCSCI test and will not be duplicated.
Clinical exam - Voluntary contraction | During enrollment, up to one week
  An SCI-specialized clinician will assess the participant in regard to the lowest area of the body that the participant is able to contract voluntarily. This data is incorporated in the ISNCSCI test and will not be duplicated.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Anderson, PhD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical System Old Brooklyn Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified set will be transferred to the Inter-University Consortium for Political and Social Research (ICPSR) for data sharing and long-term preservation.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months of end of study.
Access Criteria: Based on the ICPSR guidelines.

DOCUMENTS (1):
  • Informed Consent Form (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT05626816/ICF_001.pdf